CLINICAL TRIAL: NCT03268044
Title: The Association Between Weekend Admission and Perioperative Adverse Outcomes for Adults Undergoing Surgery: A Matched Cohort Study
Brief Title: Surgical Admission at the Weekend and 30-day Mortality in Ontario, Canada: a Matched Cohort Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, James O'Leary, Principal Investigator, The Hospital for Sick Children
Other Study IDs: 1000055744
Record Dates: First submitted 2017-08-29; First posted 2017-08-31 (Actual); Last update posted 2018-05-09 (Actual); Status verified 2018-05

CONDITIONS: Surgery
MeSH Terms: interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Weekend admission: Adults admitted to hospital at the weekend (Saturday or Sunday) and who underwent surgery
  Interventions: Other: Hospital admission and surgery
- Weekday admission: Adults admitted to hospital on a weekday (Tuesday to Thursday) and who underwent surgery
  Interventions: Other: Hospital admission and surgery

INTERVENTIONS:
Other: Hospital admission and surgery — Hospital admission and noncardiac surgery

SUMMARY:
Surgery is performed at the weekend for risk to life or limb, when mandated by clinical guidelines, or depending on resource availability. Weekend healthcare interventions have been associated with increased mortality and adverse clinical outcomes in the majority of the literature examining the weekend effect, but these findings are not consistent. Results from recent observational studies argue against a true weekend effect. Higher rates of adverse outcomes associated with hospital activity at weekends do not appear to be due to altered medical staffing as commonly hypothesized, but are thought to be in part a result of data artefact and confounding by severity or indication. For this study, we hypothesized that patients who are admitted to hospital at the weekend and require surgery have an increased risk of death compared with patients who are admitted and undergo surgery on weekdays. The primary aim was to examine whether patients who underwent surgery and were admitted at the weekend had an increased risk of 30 day all-cause mortality compared with patients who were admitted and underwent surgery on weekdays; secondary aim was to examine whether the timing of surgery (i.e., surgery on the same weekend or surgery on a subsequent weekday) for patients admitted at the weekend is associated with increased risk of 30 day all-cause mortality.

ELIGIBILITY:
Inclusion Criteria:

* any hospital admission associated with an eligible surgical procedure in the Ontario discharge abstract database
* between 2005 and 2015

Exclusion Criteria:

* cardiothoracic or cardiology therapeutic procedures
* non-surgical therapeutic interventions (e.g. dialysis)
* obstetric procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any hospital admission in Ontario, Canada, between 2005 and 2015 for noncardiac surgery.
Sampling Method: Non-Probability Sample
Enrollment: 340000 (Estimated)
Dates: Start 2016-10-18 (Actual); Primary Completion 2018-09-15 (Estimated); Study Completion 2018-09-15 (Estimated)

PRIMARY OUTCOMES:
30 day all cause mortality | 30 days from surgery
  death

CONTACTS AND LOCATIONS:
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
Study data used are housed at the Institute for Clinical Evaluative Sciences